CLINICAL TRIAL: NCT05948527
Title: Safety and Efficacy of High Flow Nasal Canula in Patients With Mild Hypercapnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R.22.12.1978.R1.R2
Record Dates: First submitted 2023-06-24; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-06

CONDITIONS: Hypercapnia
Keywords: hypercapnia; high flow nasal canula
MeSH Terms: conditions — Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- with mild Hypercapnia (Pco2 range 45-60 mmhg and power of hydrogen not less 7.30) (Experimental): with mild Hypercapnia (Pco2 range 45-60 mmhg and power of hydrogen not less 7.30) of different pulmonary disorders
  Interventions: Device: high flow nasal canula

INTERVENTIONS:
Device: high flow nasal canula — administration of high flow nasal canula at initial flow 35 liters per minute and Fio2 (fraction of inspired oxygen of 50%) with titration to reach oxygen saturation of 88-92%.

SUMMARY:
Evaluate safety and efficacy of application ( high flow nasal canula) in cases with mild hypercapnia, included 30 patients who were hospitalized in Mansoura University chest department with mild Hypercapnia (Pco2 range 45-60 mmhg and power of hydrogen not less 7.30) of different pulmonary disease categories (Chronic obstructive pulmonary disease acute exacerbation, pneumonia, Interstitial lung diseases, etc).

ELIGIBILITY:
Inclusion Criteria:

* patients with mild Hypercapnia

Exclusion Criteria:

* Excluded cases had age less than 18 years or pediatric group .
* patients with their mental state altered, confused, comatose, severe agitation or non cooperative
* Cases with moderate or severe Hypercapnia
* cases in need for immediate invasive mechanical ventilation
* cases with respiratory rate more than 35 breath per minute.
* cases with Respiratory exhaustion , fatigue , excess use of respiratory accessory muscles
* Shock , hemodynamic instability, post arrest cases,
* cases with facial trauma or severe nasal deformity,
* Patients with sleep breathing disorders or upper airway obstruction
* patients with history of home ventilation prior admission

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Arterial Blood Gases changes | 48 hours
  The primary outcome was concerned about changes in Arterial Blood Gases in first 24 h after admission and the same changes 48 h after admission.

SECONDARY OUTCOMES:
Number of participants in need for ventilation | 7 days
  Secondary outcome was concerned about need to non invasive mechanical ventilation or invasive mechanical ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
study protocol